CLINICAL TRIAL: NCT06067516
Title: Effects of Fluid Resuscitation on Capillary Refilling Time and Organ Functions in Septic Shock
Status: Completed | Type: Observational
Sponsor: Samsun University (Other)
Responsible Party: Sponsor
Other Study IDs: SUKAEK-2023 15/14
Record Dates: First submitted 2023-09-14; First posted 2023-10-05 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-06

CONDITIONS: Sepsis
Keywords: Sepsis; Fluid resuscitation; Capillary refill time; Sequential Organ Failure Assessment
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group CRT-R: If the CRT measured at T1 decreased equal to or more than 25% compared to the CRT measured at T0
  Interventions: Other: Fluid resuscitations
- Group CRT-NR: If the CRT measured at T1 decreased by less than 25% compared to the CRT measured at T0
  Interventions: Other: Fluid resuscitations

INTERVENTIONS:
Other: Fluid resuscitations — In line with the recommendations in the Surviving Sepsis Guide, fingertip capillary refill time (CRT) will be measured by applying pressure to the index finger for 15 seconds in the T1 time period after 30 mL/kg/3 hours crystalloid infusion.

SUMMARY:
Since the ultimate target of resuscitation is the microcirculation, normal microcirculatory perfusion appears to be the primary target of ideal resuscitation in septic shock patients. In septic shock patients, microcirculation of the skin may be impaired in the early period due to early sympathetic nervous system activation.

Assessment of skin perfusion has also become popular in shock resuscitation because it is easily accessible for clinical assessment. Studies in septic shock patients, showed that capillary refill time correlated with lactate levels measured at 6 hours of resuscitation and was associated with mortality. Additionally, early normalization of capillary refill time has been associated with improved survival in septic shock This study aimed to evaluate the relationship between the change in capillary filling time (microcirculation) and organ perfusion after fluid resuscitation in sepsis patients in intensive care.

DETAILED DESCRIPTION:
An aggressive approach to fluid resuscitation in patients with sepsis is recommended by international guidelines and is considered the cornerstone of treatment. This approach is based on historical concepts and the theory that septic shock is a form of hypovolemic shock characterized by tissue hypoperfusion.

Studies show that capillary refill time is a valuable method to measure the severity of acute disease both in the early and late stages. However, it remains unclear why abnormal peripheral perfusion increases morbidity and mortality. Because from a pathophysiological point of view, the main purpose of activation of the sympathetic nervous system is to maintain the perfusion of vital organs (brain, heart, lung).

The Sequential Organ Failure Assessment (SOFA) score is a simple and objective score that allows for calculation of both the number and the severity of organ dysfunction in six organ systems (respiratory, coagulatory, liver, cardiovascular, renal, and neurologic) and the score can measure individual or aggregate organ dysfunction.

This study aimed to evaluate the relationship between the change in capillary filling time (microcirculation) and SOFA score (organ perfusion) after fluid resuscitation in sepsis patients in intensive care.

After the first admission to the intensive care unit [T0 (baseline)], demographic information of the patients, source of sepsis, Sequential Organ Failure Assessment (SOFA) score, which shows the severity of the disease, Acute Physiology and Chronic Health Evaluation (APACHE II) score, additional systemic diseases, hemodynamic variables, blood gas parameters, and transthoracic echocardiogram findings will be recorded.

Capillary refill time (CRT) will be measured by applying pressure to the index finger for 15 seconds.

As recommended in the Surviving Sepsis Campaign Guidelines, after 30 mL/kg/3 hours crystalloid infusion (T1) and 24 hours (T2), Sequential Organ Failure Assessment (SOFA) score, hemodynamic variables, blood gas parameters, transthoracic echocardiogram findings and capillary refill time will be recorded again.

Patients will be divided into two groups; If the CRT measured at T1 decreased equal to or more than 25% compared to the CRT measured at T0, the patients as responders to capillary refill time (Group CRT-R); If the CRT measured at T1 decreased by less than 25% compared to the CRT measured at T0, the patients as non-responders to capillary refill time (Group CRT-NR) The effect of 30 mL/kg/3 hours crystalloid infusion on peripheral perfusion (in Group CRT-R and Group CRT-NR, which are divided into two by CRT measurement at T0 and T1 times) and the effect on the SOFA scores will be compared.

ELIGIBILITY:
Inclusion Criteria

* Over 18 years old
* Admitted to intensive care with a diagnosis of sepsis or septic shock
* Systolic blood pressure < 90 mmHg or Mean blood pressure < 65 mmHg
* Those who need vasopressor medication
* Urine output < 0.5 ml/kg/h for at least two hours
* Tachycardia (Heart rate > 100/min)
* Serum Lactate > 2 mmol/L
* Patients with central venous oxygen saturation (ScvO) < 70%

Exclusion Criteria

* Not approved by the patient or his/her guardian
* Known heart, kidney, liver failure
* The initial cause of shock is neurogenic, cardiogenic or obstructive shock.
* Pregnancy or suspected pregnancy
* Those with amputation or severe organ ischemia
* Those with peripheral artery disease
* Cannot be evaluated optimally with transthoracic echo
* Patients who died in the first 24 hours

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients admitted to intensive care due to sepsis and septic shock.
Sampling Method: Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2023-10-25 (Actual); Primary Completion 2026-01-05 (Actual); Study Completion 2026-01-05 (Actual)

PRIMARY OUTCOMES:
Sequential organ failure assessment score | up to 24 hours
  The sequential organ failure assessment score, previously known as the sepsis-related organ failure assessment score, is used to track a person's status during the stay in an intensive care unit to determine the extent of a person's organ function or rate of failure. The score is based on six different scores, one each for the respiratory, cardiovascular, hepatic, coagulation, renal and neurological systems. Each organ system is assigned a point value from 0 (normal) to 4 (high degree of dysfunction/failure). Total the Sequential organ failure assessment score ranges from 0 to 24. The Sequential organ failure assessment score is 0 to 6: mortality < 10%, 7 to 9: mortality 5 - 20%. 10 to 12: mortality 40 - 50%, 13 to 14: mortality 50 - 60%, 15: mortality > 80%, 15 to 24: mortality > 90%. The sequential organ failure assessment score changes after fluid loading (normal value sequential organ failure assessment score < 2).

SECONDARY OUTCOMES:
Stroke volume | up to 24 hours
  Stroke volume is the volume of blood pumped from the left ventricle per beat. Stroke volume is calculated using measurements of ventricle volumes from an echocardiogram and subtracting the volume of the blood in the ventricle at the end of a beat. Stroke volume change after fluid loading (normal value stroke volume 50 to 100 mL.)
Cardiac output | up to 24 hours
  Cardiac output is the amount of blood pumped by the heart minute and is the mechanism whereby blood flows around the body, especially providing blood flow to the brain and other vital organs. Cardiac output change after fluid loading (normal value stroke volume 5-6 L/min.)

OTHER OUTCOMES:
Mortality | up to 28 days
  Mortality according to capillary refill time after fluid loading in septic shock patients

CONTACTS AND LOCATIONS:
Overall Officials: OZGUR KOMURCU, 1, Principal Investigator — Samsun University
Locations (1):
- Samsun University, Samsun, Ilkadim, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jacquet-Lagreze M, Bouhamri N, Portran P, Schweizer R, Baudin F, Lilot M, Fornier W, Fellahi JL. Capillary refill time variation induced by passive leg raising predicts capillary refill time response to volume expansion. Crit Care. 2019 Aug 16;23(1):281. doi: 10.1186/s13054-019-2560-0. PMID 31420052
- [Background] Lara B, Enberg L, Ortega M, Leon P, Kripper C, Aguilera P, Kattan E, Castro R, Bakker J, Hernandez G. Capillary refill time during fluid resuscitation in patients with sepsis-related hyperlactatemia at the emergency department is related to mortality. PLoS One. 2017 Nov 27;12(11):e0188548. doi: 10.1371/journal.pone.0188548. eCollection 2017. PMID 29176794
- [Background] Brunauer A, Kokofer A, Bataar O, Gradwohl-Matis I, Dankl D, Bakker J, Dunser MW. Changes in peripheral perfusion relate to visceral organ perfusion in early septic shock: A pilot study. J Crit Care. 2016 Oct;35:105-9. doi: 10.1016/j.jcrc.2016.05.007. Epub 2016 May 12. PMID 27481743
- [Background] Monnet X, Shi R, Teboul JL. Prediction of fluid responsiveness. What's new? Ann Intensive Care. 2022 May 28;12(1):46. doi: 10.1186/s13613-022-01022-8. PMID 35633423